CLINICAL TRIAL: NCT07354620
Title: A Pilot Study on Reverse Aging (The REVERSE Study)
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: The Christ Hospital (Other)
Responsible Party: Principal Investigator, Steve Amoils, Principal Investigator, The Christ Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 24-088
Record Dates: First submitted 2025-12-11; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Aging
Keywords: Aging; Reverse Aging; Rapamycin; Biological Age; Chronological Age; Prolon
MeSH Terms: interventions — Sirolimus; Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Rapamycin Only (Experimental): 12 participants: 10 mg initial bolus dose of rapamycin followed by a weekly 6 mg rapamycin, enrolling 6 men, 6 women, with 6 ( 3 M, 3 F) who are 50-65 years; 6 ( 3 M, 3 F) who are >65 years
  Interventions: Drug: Rapamycin (Tablets)
- Prolon Diet Only (Active Comparator): 12 participants: 6 men, 6 women, with 6 (3 M, 3 F) who are 50-65 years; 6 who are >65 years Prolon® 5-day diet at 0, 1, 2, 3, 4 and 5 months;
  Interventions: Dietary Supplement: Prolon diet
- Rapamycin and Prolon Diet (Experimental): 24 participants: 10 mg initial bolus dose of rapamycin followed by a weekly 6 mg rapamycin along with Prolon 5-day diet at 0, 1, 2, 3, 4,and 5 months. : 12 men, 12 women, 12 ( 6 M, 6 F) who are 50-65 years; 12 ( 6 M, 6 F) who are >65 years.
  Interventions: Drug: Rapamycin (Tablets); Dietary Supplement: Prolon diet

INTERVENTIONS:
Drug: Rapamycin (Tablets) — 10 mg initial bolus dose of rapamycin followed by a weekly 6 mg rapamycin
  Arms: Rapamycin Only; Rapamycin and Prolon Diet
Dietary Supplement: Prolon diet — Prolon 5-day diet at 0, 1, 2, 3, 4,and 5 months
  Arms: Prolon Diet Only; Rapamycin and Prolon Diet

SUMMARY:
Aging can be defined as a time-dependent functional decline in physiological function, which may increase the vulnerability to diseases and eventually death. The question is whether aging is a normal process, or exists as an "uber-illness?" Work done by Dr Sinclair at Harvard suggests the latter. Dr. Sinclair feels people should be able to age-in-place, or even reverse age. Aging is arguably the single biggest risk factor for all acquired and chronic diseases. Delaying the aging rate by 7 years would cut the incidence of chronic disease in half! Up until know the effects of anti-aging would need longitudinal studies until death.

Now, with the advent of a 3rd generation OMIC Age clock, there is a way to assess if an intervention is changing the rate of aging and other methylation patterns associated with aging.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be healthy and of any sex, any ethnicity, and any age from 50 to 80
* "Healthy" subjects will be defined as a real-world cohort of individuals likely to utilize such an intervention
* May be on other medications if they do not conflict with rapamycin.
* All medical conditions need to be stable and well controlled.
* Willing and able to provide informed consent

Exclusion Criteria:

* Severe illnesses, for which rapamycin may cause harm. This would not be limited to but include active neoplastic or auto-immune disease. If patients have a previous history of cancer or auto-immune disease, the risks and benefits and possible adverse reactions will be discussed at time of consent
* History of organ transplant
* Any unstable medical condition that would interfere with the study
* Hepatic impairment. Note: Patients with elevated liver enzymes and low albumin, will be further screened for hepatic impairment. Elevated liver enzymes < 2x upper limit of normal will not be considered hepatic impairment.
* Renal impairment, indicated by a serum creatinine > 1.4 mg/dL
* Anemia indicated by a hemoglobin < 12 g/dL
* Platelets < 80,000/cumm,
* ANC < 1,000 / cumm
* Total WBC < 3,000/cumm
* Pregnancy or breastfeeding or woman of childbearing potential with inadequate contraception
* Unstable mental illness
* A condition where rapamycin may interfere deleteriously with a medication that is taken by a potential subject
* Currently prescribed with high dose CYP3A4 pathway medications such as verapamil > 240 mg; simvastatin >40 mg, lovastatin > 40 mg or atorvastatin > 40 mg daily. Poor GI motility as demonstrated by delayed gastric emptying on a radionucleotide isotope scan.
* Intercurrent severe infection at initiation of study drug
* Any and all other reasons that the investigator may determine that the participant is not suitable for study enrollment.
* History of or active eating disorders as deemed by PI.
* BMI lower than 18.5
* Any medication that may dangerously lower glucose while on the FMD. This will include insulin, sulfonylureas (glyburide; glipizide); Thiazolidenediones ( eg piogltazone; rosiglitazone); GLP1 drugs (semaglutide; tirzepatide);; DPP-4 inhibitors (eg sitagliptin; saxagliptin); Alpha -glucosidase inhibitors (acarbose; miglitol). Patients on SGLT2 inhibitors (empagliflozin; canagliflozin) and Metformin (glucophage) may be included in the study.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2025-02-15 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Change in Biological Age from Baseline to End of Study based on Tru Diagnostic Tru Age OMICm Age test results. | 24 weeks
  To evaluate the gradated effects of mTOR inhibition on a new OMIC methylation test that evaluates biological (vs chronological) age over a six-month period.

SECONDARY OUTCOMES:
To evaluate the effects of AMPK (AMP Kinase inhibition) on aging. Change in OMICm methylation from baseline to Week 24 based on Tru Diagnostic Tru Age OMICm Age test results. | 24 weeks
  . This will duplicate studies already done utilizing a 5 day Fasting Mimicking Diet (FMD) (Prolon) on aging. The FMD diet will be administered 6 times - at monthly intervals. Change in OMICm methylation from baseline to Week 24
Effect of weekly low-dose rapamycin on aging based on Tru Diagnostic Tru Age OMICm Age test results. | 24 weeks
  Change in OMICm methylation from baseline to Week 24
Lowering of insulin resistance based on Tru Diagnostic Tru Age OMICm Age test results. | 24 weeks
  To evaluate the combined effects of AMPK and low-dose weekly rapamycin, at lowering insulin resistance, and thereby PI3K (PI3 kinase).
Effects on insulin resistance | 24 weeks
  To stratify outcomes of the prior three outcomes based on insulin resistance. This will be monitored using a Quest Lab Insulin Resistance panel to determine if insulin resistance is a confounding variable from any of the above. Variability of results in a, b, or c based on high, low or moderate insulin resistance.
Does reversal of age improve cognition based on the Cognitive Flexibility Inventory. | 24 weeks
  Changes in the Cognitive Flexibility Inventory from baseline to week 24. Scores range from 20-140, with a higher score representing a better outcome.
Patterns based on Age based on Tru Diagnostic Tru Age OMICm Age test results. | 24 weeks
  To see if any pattern exists within age group categories. (50-65; older than age 65). Change in OMICm methylation results from baseline to Week 24 by two sub populations: ages 50-65 and ages older than age 65
Sex Difference based on Tru Diagnostic Tru Age OMICm Age test results. | 24 weeks
  Change in OMICm methylation from baseline to Week 24 by male vs female
Safety and tolerability of rapamycin and Prolon | 28 weeks
  Review of adverse reactions from baseline to Week 28

CONTACTS AND LOCATIONS:
Locations (1):
- AIM for Wellbeing, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No